CLINICAL TRIAL: NCT05298774
Title: Myoelectric Activity Following Colorectal Surgery and Return of Bowel Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: G-Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000032548
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Gastrointestinal Diseases; Ileus Paralytic; Ileus
MeSH Terms: conditions — Gastrointestinal Diseases; Ileus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Postoperative recovery with G-tech WPS (Experimental)
  Interventions: Device: G-tech WPS

INTERVENTIONS:
Device: G-tech WPS — G-tech WPS patches applied and activated within 4 hours of surgery

SUMMARY:
The purpose of the study is to determine if the myoelectrical measurements made by the G-Tech Wireless Patch System correlate with clinical markers of postoperative recovery such as passage of flatus/bowel movement, oral tolerance of diet and discharge readiness. Subsequently the data will be studied to establish which information in the signals is important in determining when to feed patients and possibly discharge them.

These pilot prospective, open clinical studies suggests that myoelectrical activity, measured on the abdominal surface with a noninvasive wireless patch system, carries predictive value in determining time to feeding and time to flatus following open abdominal surgery. Having such information in advance of clinical measures could facilitate timely interventions, be it early feeding or delaying feeding as dictated by the patient's unique recovery profile. The G-Tech Wireless Patch System would provide a unique insight into the process allowing for a tailored protocol that could improve patient satisfaction and optimize recovery. The system could also enable feedback on the impact to the overall gastrointestinal myoelectrical activity of medications, particularly opioids, used for pain management that are known to inhibit gastrointestinal function by disrupting the normal recovery patterns of colonic motility.23-25 While it remains to be seen, in addition to predicting time to flatus/bowel movement early on, the ability to continue monitoring the patient may allow one to predict onset of secondary complications, such as wound infections or anastomotic leaks, that are associated with ileus. Similarly, given the wireless noninvasive nature of the system the patients could be discharged home with the patches, whereby they would serve as a remote monitoring tool. This could be particularly useful in cases where the patients may have been discharged early and may be at a high risk for readmission. The system would then send updates/alerts to the care team for management and potentially avoid preventable readmissions.

DETAILED DESCRIPTION:
Gastrointestinal recovery after any visceral surgery is a complex dynamic process with multiple factors ranging from complexity of the surgery, degree of bowel handling and preoperative comorbidities affecting whether the recovery happens over few days, or is a slow prolonged affair lasting weeks. Delays in the gastrointestinal recovery process or ileus is accompanied by distention of the abdomen, pain, nausea, vomiting and the inability to tolerate oral feeding. Interventions to alleviate the ileus/distention include insertion or reinsertion of a nasogastric tube, instating nil per os and, if necessitated, parenteral nutrition. All of these factors contribute not only to patient discomfort, but extend length of stay (LOS), increase hospital resource utilization and thereby add to overall costs.

Clinically, the markers of gastrointestinal recovery are noted by passage of flatus, defecation and the ability to tolerate solid food without significant nausea and vomiting. Passage of stool or flatus - considered a surrogate for intestinal and anastomotic continuity - is often used as the trigger to start stepwise dietary orders with the patient's ability to tolerate each step marking their readiness for the subsequent meal. Fast-track and Enhanced Recovery After Surgery (ERAS) programs that promote early feeding in advance of these clinical markers, along with opioid sparing techniques and use of minimally invasive procedures have been shown to be safe and beneficial for many patients by demonstrating earlier recovery and shorter length of stay. However, it has also been shown that, for as many as 25% of cases, the strategy does not work as noted earlier, with the need for reinsertion of the nasogastric tube and reinstating nil per os status. In a recent study of 513 consecutive colorectal patients who were on an ERAS protocol, 128 patients (24.7%) needed postoperative reinsertion of nasogastric tube at the 3.9±2.9 postoperative day. This suggests that, while early postoperative feeding is beneficial to patients in whom recovery is on track, it does not work in cases where patients are not ready for it.

At present, there is no reliable measurement that can predict gastrointestinal recovery/diet readiness for patients in advance of these clinical markers that may allow for interventions or fast-track programs to facilitate timely recovery. Auscultation for return of bowel sounds, long part of the standard of care, is controversial in its usefulness to indicate recovery. Bowel sounds have shown to have poor correlation with flatus/defecation and have proved unsuccessful in guiding diet interventions.

Smooth muscle electrical activity on the other hand is directly related to gastrointestinal function and motility. Researchers have previously shown a 1:1 correlation between electrical and mechanical (contractile) events in the colon with internally placed electrode-strain gauge force transducers. Electrical activity in the colon has been reported across a wide range of frequencies ranging from 0 to 40 cycles per min (cpm)). Condon et. al have documented the progressive return of colonic electrical related to resolution of postoperative ileus and clinical recovery following surgery. These measurements have been performed using electrodes placed internally during surgery, a major impediment towards broader use of such technology.

G-Tech Medical has developed a noninvasive wireless patch system that measures electrical activity from the gastrointestinal smooth muscles on the abdominal surface. This technology has been studied as part of several non-significant risk IRB approved studies in both adults and pediatric populations to evaluate the patterns of gastrointestinal myoelectrical signals following surgery. The studies demonstrate that signals measured by the G-Tech Wireless patches correlate with clinical markers of postoperative recovery such as time to feeding and time to flatus following pancreaticoduodenectomy and general abdominal surgeries respectively. The study in patients undergoing pancreaticoduodenectomy procedures was conducted in collaboration with researchers at Stanford University. The study demonstrated that measurement of gastric activity beginning immediately after pancreaticoduodenectomy with the G-Tech Wireless Patch System, based on the measured spectral peak near 3 cpm, could distinguish patients with shorter or longer times to diet readiness. The study demonstrated the potential utility of the G-Tech Patch System in providing objective data to identify patients who are progressing as well as, or better than expected, and those who are at risk for delayed gastric emptying. In another open, prospective study, researchers examined the use of the G-Tech Wireless Patch System in predicting time to first flatus by looking at colonic myoelectrical activity following general abdominal surgeries.21 Patients with early flatus had stronger early colonic activity than patients with late flatus. At 36 h post-surgery, a linear fit of time to flatus vs cumulative colonic myoelectrical activity predicted first flatus as much as 5 days (± 22 h) before occurrence.

These pilot prospective, open clinical studies suggests that myoelectrical activity, measured on the abdominal surface with a noninvasive wireless patch system, carries predictive value in determining time to feeding and time to flatus following open abdominal surgery. Having such information in advance of clinical measures could facilitate timely interventions, be it early feeding or delaying feeding as dictated by the patient's unique recovery profile. The G-Tech Wireless Patch System would provide a unique insight into the process allowing for a tailored protocol that could improve patient satisfaction and optimize recovery. The system could also enable feedback on the impact to the overall gastrointestinal myoelectrical activity of medications, particularly opioids, used for pain management that are known to inhibit gastrointestinal function by disrupting the normal recovery patterns of colonic motility. While it remains to be seen, in addition to predicting time to flatus/bowel movement early on, the ability to continue monitoring the patient may allow one to predict onset of secondary complications, such as wound infections or anastomotic leaks, that are associated with ileus. Similarly, given the wireless noninvasive nature of the system the patients could be discharged home with the patches, whereby they would serve as a remote monitoring tool. This could be particularly useful in cases where the patients may have been discharged early and may be at a high risk for readmission. The system would then send updates/alerts to the care team for management and potentially avoid preventable readmissions.

The purpose of the Phase 1 study is to determine if the myoelectrical measurements made by the G-Tech Wireless Patch System correlate with clinical markers of postoperative recovery such as passage of flatus/bowel movement, oral tolerance of diet and discharge readiness. Subsequently the data will be studied to establish which information in the signals is important in determining when to feed patients and possibly discharge them.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. Eighteen (18) years of age or older
3. Subject is willing and able to follow all study requirements
4. Subject has undergone or will undergo a laparoscopic or open colorectal surgery with resection and anastomosis

Exclusion Criteria:

1. Subject is pregnant or suspects pregnancy.
2. Known allergy to medical grade adhesive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Postoperative Recovery With G-tech WPS: Patients had G-tech WPS patches applied and activated within 4 hours of surgery
Period: Overall Study
Arm/Group | Postoperative Recovery With G-tech WPS
Started | 77
Completed | 68
Not Completed | 9
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 3
Not completed — Screen failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Postoperative Recovery With G-tech WPS
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.42 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 70
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 67
  More than one race | 1
  Unknown or Not Reported | 1
Height [Mean (Standard Deviation); unit: cm] | 170.27 (10.60)
Weight [Mean (Standard Deviation); unit: kg] | 79.88 (19.43)

OUTCOME MEASURES:

1. Primary Outcome: GI Functional Recovery
Description: Time to return of flatus or bowel movement after colorectal surgery
Time Frame: 30 days after index surgery
Population: Of the 77 participants assigned to the arm, 7 did not receive the G-tech WPS patches after enrollment, and outcome data was not recorded for 3 additional participants. Therefore, 67 participants were included in the analysis population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Postoperative Recovery With G-tech WPS
Number analyzed (Participants) | 67
hours | 47.94 (30.78)

2. Secondary Outcome: Postoperative Ileus
Description: Occurrence of postoperative ileus after colorectal surgery
Time Frame: 30 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Postoperative Recovery With G-tech WPS
Number analyzed (Participants) | 77
Participants | 6

3. Secondary Outcome: Readmission With Ileus
Description: Occurrence of readmission with postoperative ileus after colorectal surgery
Time Frame: 30 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Postoperative Recovery With G-tech WPS
Number analyzed (Participants) | 77
Participants | 0

ADVERSE EVENTS:
Time Frame: 14 days of follow-up after index surgery
Arm/Group | Postoperative Recovery With G-tech WPS
All-Cause Mortality (participants affected / at risk) | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77
Other Adverse Events (participants affected / at risk) | 0/77

LIMITATIONS AND CAVEATS:
The study is limited by a short follow-up duration restricted to in-patient settings and aligning myoelectric readings with clinical symptoms is under-powered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT05298774/Prot_SAP_ICF_001.pdf